CLINICAL TRIAL: NCT01505036
Title: Randomized, Multi-center, Open-label, Parallel Group Study to Evaluate the Effect of the Smart Care-diabetes Management System on Subjects With Diabetes
Brief Title: Study to Evaluate the Effect of the Smart Care-diabetes Management System on Subjects With Diabetes
Acronym: SMARTCARE_DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SK Telecom Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMARTCARE_DM
Record Dates: First submitted 2011-07-19; First posted 2012-01-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; smart-care; U-health care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMARTCARE service (Experimental): U-Health service
  Interventions: Other: SMARTCARE service
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: SMARTCARE service — U-Healthcare service
  Other Names: U-Healthcare
  Arms: SMARTCARE service

SUMMARY:
SMARTCARE-diabetes management system' to evaluate the long-term effects on patients with diabetes.

DETAILED DESCRIPTION:
Primary Outcome Measure: To see if there's any change in HbA1C at Visit 6 (12M) compared Visit 2 (baseline) within each group and between the two groups.

All statistical analysis will progress through the SAS (Version 9.1). statistical test's significance level is 0.05. The principle is two-sided test.

Secondary Outcome Measures :

To see if there's any change in HbA1C at each Visit (Visit 3 - Visit 6) compared Visit 2 (baseline) within each group and between the two groups.

Add a Secondary Outcome Measure:

Treatment satisfaction (DTSQ, Diabetes Treatment Satisfaction Questionnaire): To see if there's any change in treatment satisfaction scores compared Visit 2 (baseline) within each group and between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. At least 1 year after being diagnosed with Type 2 diabetes
3. 7.0% ≤ HbA1c ≤ 10.0%
4. Agreed to participate voluntarily in the study

Exclusion Criteria:

1. Severe chronic disease
2. Diabetes mellitus complications
3. Severe renal disease; Serum creatinin > 1.5(men), > 1.4 (women)
4. Severe liver disease or AST, ALT ≥ 2.5 x ULN
5. Known not to be taking medication reliably 3 months before the screening visit
6. Insulin pump user
7. Being registered for other clinical research or are planning to participate in other clinical researches during this study
8. Pregnant woman
9. Illiterate
10. Being assessed irrelevant by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of patients who attain,Hemoglobin A1C ≤ 7.0% and Blood pressure ≤ 130/80 and LDL-Cholesterol ≤ 100 or LDL-Cholesterol ≤ 70, all at 12 months. | 0 to 12 months
  Rate of patients who attain, Hemoglobin A1C ≤ 7.0% and Blood pressure ≤ 130/80 and and LDL-Cholesterol ≤ 100 or LDL-Cholesterol ≤ 70, all at 12 months.

SECONDARY OUTCOMES:
Change in Hemoglobin A1C at visit 3,4,6 from baseline | 0 to 12 months
  Change in Hemoglobin A1C at Visit3,4,6 from baseline. Reduce Hemoglobin A1c after study
change in QOL(Quality of life) | 0 to 12 months
  Change in QOL(Quality of life) at Visit 6 from baseline.
Treatment satisfaction(DTSQ, Diabetes Treatment Satisfaction Questionnaire) | 0 to 12 months
  change in Treatment satisfaction(DTSQ, Diabetes Treatment Satisfaction Questionnaire) at Visit 6 from baseline.
Changes in lipid profile at Visit 4 and 6 from baseline. | 0 to 12 months
  Changes in lipid profile at visit 4 and 6 from baseline. Reduction of lipid profile
Changes in body weight | 0 to 12 months
  Changes in body weight at each visit(visit 3,4,5,6) from baseline during 12 months. Reduction of body weight
Changes in Waist Circumference(WC) | 0 to 12 months
  Changes in Waist Circumference(WC) at each visit(visit 3,4,5,6) from baseline during 12 months.
  Reduction of Waist Circumference(WC)
Changes in Blood Pressure | 0 to 12 months
  Changes in Blood Pressure at each visit(visit 3,4,5,6) from baseline during 12 months.
  Changes in mean Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: kun-ho YOON, professor, Principal Investigator — Seoul St. Mary's Hospital; sung-woo PARK, Professor, Principal Investigator — Kanbuk Samsung Medical Center; Jung-yeol PARK, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Medicrostar, Seoul, South Korea